CLINICAL TRIAL: NCT05939752
Title: Cardiovascular Complications of Ibrutinib Therapy: a Single-center Cohort Study
Brief Title: Cardiovascular Complications of Ibrutinib Therapy
Acronym: CACIS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ROBERT AOI 2022
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Ibrutinib Treatment
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Patients with an indication for ibrutinib treatment for hematologic reasons
  Interventions: Other: ophthalmological examination; Biological: blood test

INTERVENTIONS:
Other: ophthalmological examination — OCT-retinal angiography At inclusion, 3 months and 6 months
Biological: blood test — a 2-mL tube of blood will be taken to test for blood markers predisposing to cardiovascular complications.
  At inclusion

SUMMARY:
Ibrutinib, the first BTK inhibitor (BTKI) to be approved, improves progression-free survival (PFS) and overall survival (OS) over alternative therapies in relapsed/refractory and treatment-naive chronic lymphocytic leukemia (CLL). Ibrutinib has also been found to be effective in mantle cell lymphoma, Waldenström's macroglobulinemia and marginal zone lymphoma. However, ibrutinib treatment is associated with an increased risk of atrial fibrillation (AF), with an estimated 2-year AF rate of 16% in patients treated with ibrutinib during a median follow-up of 28 months. In most studies, AF was identified by reports as a treatment-related adverse event, and systematic screening for AF was not performed. As AF is often paroxysmal, the more intensive the screening, the higher the incidence. In a prospective cohort study of 53 patients treated with ibrutinib for CLL, patients were monitored by pulse palpation and ECG every 3 months. The cumulative incidence rate of ibrutinib-associated AF was 23% at 12 months and 38% at 2 years. The management of ibrutinib-associated AF is challenging due to difficulties in balancing the benefits of anticoagulation to mitigate the risk of stroke and the bleeding risk associated with ibrutinib. AF is a frequent reason for discontinuation of ibrutinib therapy, and can result in significant morbidity.

In addition to this arrhythmogenic effect, ibrutinib is also significantly associated with the onset or worsening of arterial hypertension. Finally, an increased risk of serious ventricular rhythm disorders has also been suggested by pharmacovigilance databases, but not yet confirmed by prospective clinical studies.

The study proposes a comprehensive cardiovascular approach, at baseline and during follow-up of patients on Ibrutinib, using innovative markers to anticipate patients most at risk of developing these cardiovascular effects, but also to detect them as early as possible in order to avoid the complications they may generate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for ibrutinib treatment for hematologic reasons
* Patients aged 18 and over
* Patients who have given their free, written and informed consent to this study after being informed (or by the patient's representative if the patient is unable to express his or her consent).

Exclusion Criteria:

* Person not affiliated to national health insurance
* Patient under legal protection (curatorship, guardianship)
* Patient subject to a safeguard of justice measure
* Pregnant, parturient or breast-feeding women
* Previous treatment with ibrutinib
* Follow-up planned in another center
* History of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified by a doctor working in the hematology department of Dijon University Hospital during his or her regular medical check-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
rate of patients developing atrial fibrillation (AF) | 12 months after introduction of ibrutinib
  Compare the values of selected biomarkers between patients who have developed AF and patients without AF

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France